CLINICAL TRIAL: NCT06236711
Title: A Feasibility Study of Transcranial Direct Current Stimulation (tDCS) as an Adjunctive Treatment for Treatment Resistant Depression (TRD) in Hospitalized Patients
Brief Title: Transcranial Direct Current Stimulation (tDCS) as an Adjunctive Treatment for Treatment Resistant Depression (TRD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Lapid, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-003274
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- tDCS interventional arm (Experimental): Participants will receive a 30-minute tDCS treatments at 2 mA twice daily over the course of 5 days.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS is a form of noninvasive transcranial stimulation of the brain by delivering low-intensity electrical current to the scalp through two electrodes. The Soterix Medical 1×1 Low Intensity Transcranial DC Stimulator Model 1300A (Soterix Medical, Inc., New York, NY, USA) device will be used in the study. The tDCS device is comprised of a small battery-operated control box that delivers the current through electrodes placed on the scalp, held in place by elastic bands or head straps and worn over the forehead like a headband.

SUMMARY:
The researchers are trying to test the feasibility and acceptability of using transcranial Direct Current Stimulation (tDCS) in hospitalized adult patients with Treatment Resistant Depression (TRD), assess for any preliminary effect on depressive and cognitive symptoms, and explore the utility of biomarkers to assess response to tDCS.

DETAILED DESCRIPTION:
In this feasibility study the researchers propose to conduct a 5-day tDCS treatment protocol in hospitalized adult patients with TRD, with each treatment session lasting for 30 minutes, delivered twice daily, for a total of 10 stimulations over 5 days. Before and after the 5-day tDCS treatment protocol, assessments will include Montgomery-Asberg Depression Rating Scale (MADRS) to measure depressive symptoms, Snaith-Hamilton Pleasure Scale (SHAPS) to measure anhedonia, Stroop Test to measure memory and executive function, Revised Hopkins Verbal Learning Test (HVLT-R) to test verbal learning and memory, and Digital Symbol Coding Test (DSCT) to measure working memory. Electroencephalography (EEG) for objective electrophysiologic data will also be collected before and after tDCS. A wireless EEG unit (CGX, Cognionic, Inc.) will be used to collect EEG and peak alpha frequency (PAF) as potential target engagement marker for tDCS. The PAF measures the highest magnitude within the alpha range of brain oscillations, thought to reflect cognitive performance. Other potential predictors of treatment response measures collected at baseline include Adverse Childhood Experiences (ACE), premorbid intelligence quotient (pIQ), Wide Range Achievement Reading Test (WRART), and Socioeconomic Status (SES).

ELIGIBILITY:
Inclusion Criteria

* 18 years and older
* Clinical diagnosis of treatment-resistant depression (defined as depression that does not remit following two or more treatment attempts of an adequate dose and duration of a minimum duration of 4 weeks)
* Hospitalized in psychiatric units
* Voluntary admission status
* Moderate or severe depression, defined by PHQ-9 ≥ 15
* Ability to provide informed consent
* Ability to adhere to protocol

Exclusion Criteria

* Bipolar disorder
* Active primary psychotic or substance use disorders (except nicotine dependence) within the past year
* Any active neurological condition (including seizure disorder, traumatic brain injury, stroke)
* Contraindications to tDCS (including pacemaker, metallic implants in the head or neck [except orthodontic hardware], skin disease causing irritation)
* Current pregnancy or positive urine pregnancy test (clinical)
* Any neuromodulation therapy (including ECT, rTMS, DBS, VNS, TES) within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcome | through study completion, an average of 2 weeks
  Defined as 70% of eligible patients choosing to enroll in the study. Other feasibility parameters will include willingness of clinicians to refer and help recruit patients, number of eligible participants, willingness of participants to enroll, retention of patients, and completeness of data collection.
Acceptability outcome | through study completion, an average of 2 weeks
  Defined as 80% of study participants completing 80% of the 10-session tDCS treatment protocol. Investigators will also ask participants about their satisfaction, perceptions, and experiences with the tDCS treatments. Other acceptability parameters will include rates of adherence to tDCS protocol, dropout rates and reasons for non-completion.
Tolerability outcome | through study completion, an average of 2 weeks
  Defined as an overall tolerability rating of "very tolerable." This will be a self-report based on a global question "Considering all aspects of your experience, how would you rate the overall tolerability of the tDCS intervention?" The response options are: very tolerable, somewhat tolerable, neutral, somewhat intolerable, and very intolerable. Other tolerability parameters will include the tDCS adverse effects questionnaire.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | baseline, 2 weeks
  Measure of depressive symptoms. Response is defined by a 50% or more reduction in MADRS score. The MADRS has 10-items which are based on mood symptoms. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Change in Snaith-Hamilton Pleasure Scale (SHAPS) | baseline, 2 weeks
  Measure of anhedonia. The SHAPS has 14-items which are based on pleasure symptoms. Each item is scored 1 (definitely agree) to 4 (definitely disagree) with overall score ranges from 14 (experience high pleasure) to 56 (experience low pleasure)
Change in Stroop Test | baseline, 2 weeks
  Measure of measure memory and executive function. Reaction time (in seconds) in the different conditions of the task (reading the non-conflicting condition, reading the conflicting condition)
Change in Revised Hopkins Verbal Learning Test (HVLT-R) | baseline, 2 weeks
  Measure of verbal learning and memory. The HVLT-R has 12-items which are based on memory score. Total recall score (range from 0 to 36). The higher the score indicates better short-term memory, lowers scores indicates worse short-term memory.
Change in Digital Symbol Coding Test (DSCT) | baseline, 2 weeks
  Measure of working memory. The DSST involves a key consisting of the numbers 1-9, each paired with a unique, easy to draw symbol. Below the key are a series of numbers that 1-9 in random order and repeated several times, that are to be filled in the corresponding symbol for each number. One point is given for each correct response. Total scores range from 0-9, lower scores indicate worse memory; higher scores indicate better memory.
Change in Peak alpha frequency (PAF) | baseline, 2 weeks
  EEG measure of the highest magnitude within the alpha range of brain oscillations, thought to reflect cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Lapid, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li JW, Ren C, Pazdernik VK, Kung S, Basso MR, Croarkin PE, Aaron B, Anderson AM, Caves CA, Hemm MN, Holland AL, Hoth CR, Jazdzewski EA, Kabristante E, Kandimalla M, Mickle CB, Min HK, Ozger C, Parsons JM, Sheldon RL, Skime MK, St Louis EK, Varatharajah Y, Wagh N, Welker KM, Williams SM, Worrell GA, Lapid MI. Transcranial direct current simulation as an adjunctive treatment for treatment-resistant depression in hospitalized patients: A feasibility study protocol. PLoS One. 2025 Jun 10;20(6):e0324808. doi: 10.1371/journal.pone.0324808. eCollection 2025. PMID 40493630
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials